CLINICAL TRIAL: NCT01067157
Title: Long-term Effects of Lifestyle Intervention in Obesity and Genetic Influence in Children - LOGIC-Study
Brief Title: Long-term Effects of Lifestyle Intervention in Obesity and Genetic Influence
Acronym: LOGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Rehabilitation clinic Schönsicht, 83471 Berchtesgaden (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LOGIC
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Obesity; Cardiovascular Risk
Keywords: Obesity; overweight; childhood; adolescence; inpatient therapy; lifestyle intervention; cardiovascular risk; gene-lifestyle-interaction; Obesity and associated cardiovascular risk in childhood and adolescence,; health behaviour
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Other = Lifestyle intervention
  A: Medical examination before and after inpatient therapy (clinic staff), questionnaires.
  Further medical examination and questionnaires after 6 months, 1, 2, 5 and 10 years at home by pediatrics or general practitioner.
  The lifestyle intervention includes an age-specific diet (1200-1800 kcal/d), 11 h/wk physical activity (walking, swimming, sports) and behavioural therapy.
  Interventions: Behavioral: LOGIC

INTERVENTIONS:
Behavioral: LOGIC — Experimental group:
  Diet (1200-1800 kcal/d), Exercise: 11 h/wk physical activity, Behavioural therapy (group training, 1-3h/wk individualized personal instructions, 2 h parents work)

SUMMARY:
The purpose of the study is to determine the genetic influence on short-, middle- and longterm effects of an inpatient lifestyle therapy program in overweight and obese children and adolescents.

DETAILED DESCRIPTION:
In Germany, as in other countries, overweight and obesity affects a growing number of children and adolescents. Obesity-related diseases such as arterial hypertension, disorders of glucose and lipid metabolism and an increase in inflammation markers are associated with higher morbidity and mortality in early life, therefore effective therapy concepts are needed.

The aim of this study is to evaluate the effects of a 4-6 week inpatient obesity lifestyle therapy program over 10 years and the genetic influence on the short-, middle- and longterm outcome.

The lifestyle intervention consists of physical exercise, nutrition education and behaviour therapy based on the criterions developed by the German Obesity Group (degree of weight reduction, improvement of comorbidity and health behaviour, minimising of side effects).

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese children (BMI >90th percentile for age and gender), who obtained an inpatient lifestyle intervention in the participating clinic.
* Children with written consent from their parents and the acceptance of a 10-year follow-up.

Exclusion Criteria:

* Children without written consent from their parents.
* Children with monogenetic diseases with influence on obesity (e.g. Prader-Willi-Syndrome) or with secondary obesity.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Influence of gene variants in FTO, MC4R and TMEM-18 on reduction of overweight and obesity measured by standard deviation score Body Mass Index (sds-BMI) | 16 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, Prof. M.D., Study Chair — Department of Medicine, Division of Prevention, Rehabilitation and Sports Medicine, Technical University Munich, Germany
Locations (1):
- Department of Medicine, Division of Prevention, Rehabilitation and Sports Medicine, Technical University Munich, Germany, Munich, Bavaria, Germany

REFERENCES:
- [Background] Reinehr T, de Sousa G, Toschke AM, Andler W. Long-term follow-up of cardiovascular disease risk factors in children after an obesity intervention. Am J Clin Nutr. 2006 Sep;84(3):490-6. doi: 10.1093/ajcn/84.3.490. PMID 16960161
- [Background] Baker JL, Olsen LW, Sorensen TI. Childhood body-mass index and the risk of coronary heart disease in adulthood. N Engl J Med. 2007 Dec 6;357(23):2329-37. doi: 10.1056/NEJMoa072515. PMID 18057335
- [Background] Bibbins-Domingo K, Coxson P, Pletcher MJ, Lightwood J, Goldman L. Adolescent overweight and future adult coronary heart disease. N Engl J Med. 2007 Dec 6;357(23):2371-9. doi: 10.1056/NEJMsa073166. PMID 18057339
- [Background] Owen CG, Whincup PH, Orfei L, Chou QA, Rudnicka AR, Wathern AK, Kaye SJ, Eriksson JG, Osmond C, Cook DG. Is body mass index before middle age related to coronary heart disease risk in later life? Evidence from observational studies. Int J Obes (Lond). 2009 Aug;33(8):866-77. doi: 10.1038/ijo.2009.102. Epub 2009 Jun 9. PMID 19506565
- [Background] Birch LL, Ventura AK. Preventing childhood obesity: what works? Int J Obes (Lond). 2009 Apr;33 Suppl 1:S74-81. doi: 10.1038/ijo.2009.22. PMID 19363514
- [Background] Daniels SR, Arnett DK, Eckel RH, Gidding SS, Hayman LL, Kumanyika S, Robinson TN, Scott BJ, St Jeor S, Williams CL. Overweight in children and adolescents: pathophysiology, consequences, prevention, and treatment. Circulation. 2005 Apr 19;111(15):1999-2012. doi: 10.1161/01.CIR.0000161369.71722.10. PMID 15837955
- [Background] McCall A, Raj R. Exercise for prevention of obesity and diabetes in children and adolescents. Clin Sports Med. 2009 Jul;28(3):393-421. doi: 10.1016/j.csm.2009.03.001. PMID 19505623
- [Derived] Siegrist M, Heitkamp M, Braun I, Vogg N, Haller B, Langhof H, Koenig W, Halle M. Changes of omentin-1 and chemerin during 4 weeks of lifestyle intervention and 1 year follow-up in children with obesity. Clin Nutr. 2021 Nov;40(11):5648-5654. doi: 10.1016/j.clnu.2021.09.042. Epub 2021 Oct 8. PMID 34666255
- [Derived] Rank M, Siegrist M, Wilks DC, Langhof H, Wolfarth B, Haller B, Koenig W, Halle M. The cardio-metabolic risk of moderate and severe obesity in children and adolescents. J Pediatr. 2013 Jul;163(1):137-42. doi: 10.1016/j.jpeds.2013.01.020. Epub 2013 Feb 20. PMID 23434121
- [Derived] Rank M, Siegrist M, Wilks DC, Haller B, Wolfarth B, Langhof H, Halle M. Long-term effects of an inpatient weight-loss program in obese children and the role of genetic predisposition-rationale and design of the LOGIC-trial. BMC Pediatr. 2012 Mar 19;12:30. doi: 10.1186/1471-2431-12-30. PMID 22429873
- See also: Related Info — http://www.sport.med.tum.de
- See also: Related Info — http://www.klinikschoensicht.de